CLINICAL TRIAL: NCT04039555
Title: Clinical Study to Compare the Efficacy of 1 Series of 2 Treatment Sessions With Erbium-Yag Laser or CO2RE Intimate Laser vs Sham (Sham Treatment) for Vulvovaginal Atrophy (Dryness and / or Dyspareunia)
Brief Title: Clinical Study to Compare the Efficacy of Erbium-Yag Laser or CO2RE Intimate Laser With Sham (COER)
Acronym: COER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Palacios (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COER
Record Dates: First submitted 2019-04-22; First posted 2019-07-31 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Vaginal Atrophy
MeSH Terms: interventions — Lasers, Solid-State

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: It is a single blind study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Arm - CO2 intimate (Active Comparator): Patients will receive 2 sessions of CO2 laser treatment, spaced 4 to 6 weeks apart
  Interventions: Device: CO2 intimate
- Active Arm - Erbium-yag (Active Comparator): Patients will receive 2 sessions of Erbium-Yag laser treatment, spaced 4 to 6 weeks apart
  Interventions: Device: Erbium-yag
- Sham Arm (Sham Comparator): Patients will receive 2 sessions of Erbium-Yag laser or CO2 laser treatment with non-therapeutic energy, spaced between 4 and 6 weeks apart
  Interventions: Device: CO2 intimate or Erbium-yag

INTERVENTIONS:
Device: CO2 intimate — Two sessions with CO2 intimate laser for vaginal symptoms treatment
  Arms: Active Arm - CO2 intimate
Device: Erbium-yag — Two sessions with Erbium-yag laser for vaginal symptoms treatment
  Arms: Active Arm - Erbium-yag
Device: CO2 intimate or Erbium-yag — Two sessions of one of the two lasers with no therapeuthical energy
  Arms: Sham Arm

SUMMARY:
This trial compares the efficacy of two different laser treatments for vaginal atrophy symptoms between them and with sham treatment. Patients will be randomized to one of the two lasers or sham treatment.

DETAILED DESCRIPTION:
Patients over 45 years of age with one or more AVV symptoms who wish to participate in the study will be included, 2 laser sessions spaced one of another 4-6 weeks, and final tracking visit 4-6 weeks of the last laser session.

Each patient shall be randomly assigned an arm of tto, with laser CO2, or laser Erbium, or sham group

ELIGIBILITY:
Inclusion Criteria:

* Women older than 45 years with at least one year of amenorrhea and at least one symptom of vulvovaginal atrophy of moderate and / or severe intensity.

Exclusion Criteria:

* Hormone treatment in the last three months for vulvovaginal atrophy
* Treatment with vaginal moisturizers in the last week for vulvovaginal atrophy
* Laser treatment in the last 12 months.
* Acute and recurrent infections of the urinary tract in the last 3 months.
* Acute genital infections
* Vaginal prolapse
* Alterations in the area to be treated, such as lacerations, abrasions or ulcers (time of resolution at medical discretion)
* Chronic decompensated noncommunicable diseases
* Women who are pregnant or have given birth in the last 3 months

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 136 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Comparation of 1 series of 2 treatment sessions with Erbium-Yag or intimate CO2RE vs Sham for the symptoms of vulvovaginal atrophy | Visit 1(Day 0), visit 2(5 +/-1 weeks), visit 3(10 +/-1 weeks)
  Analyzing the differences in % the cytological maturity index, changes in the intensity of symptoms and PH range of normality (3,5- 4.5).

SECONDARY OUTCOMES:
Differences between CO2RE and Erbium-Yag | Visit 1(Day 0), visit 2(5 +/-1 weeks), visit 3(10 +/-1 weeks)
  Analyzing the differences in % the cytological maturity index, changes in the intensity of symptoms and PH range of normality (3,5- 4.5).
Changes in the Vulvar and Vaginal Health Index (VVHI) | Visit 1(Day 0), visit 2(5 +/-1 weeks), visit 3(10 +/-1 weeks)
  Analyzing the information registered in the visits performed

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Palacios, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No